CLINICAL TRIAL: NCT00939796
Title: A Clinical Study of the Acclarent Tympanostomy Tube Delivery System For the Treatment of Patients Requiring Tympanostomy Tube Insertion for Otitis Media (inVENT)
Brief Title: Clinical Study of the Tympanostomy Tube Delivery System
Acronym: inVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005005
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tympanostomy Tube Delivery System (TTDS) (Experimental): Tympanostomy tube placement with Acclarent tube delivery system
  Interventions: Device: Acclarent Tympanostomy Tube Delivery System

INTERVENTIONS:
Device: Acclarent Tympanostomy Tube Delivery System — A device which provides a means to create a myringotomy with insertion of a proloaded tympanostomy tube (TT) for placement of the TT in patients indicated for such treatment for Otitis Media

SUMMARY:
The objective of this investigational study is to evaluate the safety and performance of the Acclarent Tympanostomy Tube Delivery System (TTDS) for the placement of the Tympanostomy Tube [TT(s)] in patients indicated for such treatment for chronic otitis media with effusion (OME) or recurrent acute otitis media (AOM).

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo bilateral or unilateral tympanostomy tube insertion.
2. Either male or female

Exclusion Criteria:

1. History of sensitivity or reaction to anesthesia chosen for the procedure
2. Markedly atrophic, mono- or bimeric, severely retracted, atelectatic or perforated tympanic membrane
3. Otitis externa
4. Active acute otitis media
5. Otitis media pathology
6. Stenosed ear canal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Syms, III, MD, Principal Investigator — Ear Medical Group; Charles Wilson, MD, Principal Investigator — Bay Area ENT
Locations (2):
- United States (2):
  - Bay Area ENT, Biloxi, Mississippi
  - Ear Medical Group, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients presenting to the clinical practice and for whom tympanostomy tube (TT) insertion was recommended were offered the opportunity to participate in the study. Recruitment period was May-June 2009.
Pre-assignment Details: Investigators treated a minimum of 1 subject (or 2 ears) as lead-in procedures prior to enrolling test cohort. 3 lead-in subjects were enrolled and were required to meet the same eligibility criteria and protocol-required procedures as the test cohort. Lead-in efficacy data have been separately analyzed. 13 subjects enrolled in the test cohort.
Period: Overall Study
Arm/Group | Tympanostomy Tube Delivery System (TTDS)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tympanostomy Tube Delivery System (TTDS)
Number analyzed (Participants) | 16
Age, Customized [Number; unit: participants]
  <=5 years | 14
  >5 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Device Success
Description: Successful deployment of the tube in each indicated ear using the TTDS. Evaluated for test cohort subjects only (not lead-in subjects).
Time Frame: At procedure visit
Population: All TTDS devices attempted
Measure: Number; unit: devices
Units Other Than Participants: devices
Arm/Group | Tympanostomy Tube Delivery System (TTDS)
Number analyzed (Participants) | 13
Number analyzed (devices) | 26
devices | 21 [xx.x to xx.x]

2. Secondary Outcome: Cross-Over to Manual Myringotomy and Tube Placement
Description: Conversion of the procedure from Tympanostomy Tube Delivery System to manual myringotomy and tube placement. Evaluated for test cohort subjects only (not lead-in subjects). Decision to convert to a manual myringotomy and tube placement procedure occurs at the conclusion of the Tube Delivery System procedure.
Time Frame: at procedure visit
Measure: Number; unit: number of ears
Units Other Than Participants: ears attempted
Arm/Group | Tympanostomy Tube Delivery System (TTDS)
Number analyzed (Participants) | 13
Number analyzed (ears attempted) | 24
number of ears | 3 [xx.x to xx.x]

3. Secondary Outcome: Tube Retention
Description: Presence of the Tympanostomy Tube across the tympanic membrane at two weeks post-procedure. Evaluated for test cohort subjects only (not lead-in subjects).
Time Frame: two weeks post-procedure
Measure: Number; unit: retained tubes
Units Other Than Participants: retained tubes
Arm/Group | Tympanostomy Tube Delivery System (TTDS)
Number analyzed (Participants) | 13
Number analyzed (retained tubes) | 24
retained tubes | 24 [xx.x to xx.x]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Tympanostomy Tube Delivery System (TTDS)
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanostomy Tube Delivery System (TTDS) (N=16)
tympanic membrane perforation (Ear and labyrinth disorders) | 2 (2) — In the Lead-In cohort: Unintended TM perforations occurred in 2 of 6 ears recorded as non-serious device-related adverse events, with no sequelae. There were no SAEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days